CLINICAL TRIAL: NCT01490814
Title: A Controlled, Prospective, Non-Inferiority, Parallel-Group, Randomised, Interventional, Open, Blinded Outcome Assessment (PROBE-Design), Multi-centre Trial, Comparing Efficacy and Safety of Isolation of the PVs With a Cryoballoon Catheter vs a Radiofrequency Ablation With a ThermoCool Catheter in Patients With PAF
Brief Title: FIRE AND ICE: Comparative Study of Two Ablation Procedures in Patients With Atrial Fibrillation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medtronic Atrial Fibrillation Solutions (Industry)
Collaborators: Medtronic (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FI-123
Record Dates: First submitted 2011-12-06; First posted 2011-12-13 (Estimated); Results first posted 2018-11-02 (Actual); Last update posted 2018-11-02 (Actual); Status verified 2018-03

CONDITIONS: Symptomatic Paroxysmal Atrial Fibrillation (PAF)
Keywords: PAF; two episodes within the last twelve months one episode documented; Documented treatment failure of at least one antiarrhythmic; drug AAD Type I or III including β-blocker and AAD intolerance

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Cryoballoon ablation (Active Comparator)
  Interventions: Procedure: Electrical isolation of the pulmonary veins
- Radiofrequency ablation (Active Comparator)
  Interventions: Procedure: Electrical isolation of pulmonary veins

INTERVENTIONS:
Procedure: Electrical isolation of the pulmonary veins — Device: ArcticFront® Cardiac CryoAblation Catheter System with the FlexCath Steerable Sheath or ArcticFront® Advance Cardiac CryoAblation Catheter System with the FlexCath Steerable Sheath or any future development generations of this product line, provided they are CE marked and the centre has the experience of at least 10 procedures before including a patient into the study.
  Arms: Cryoballoon ablation
Procedure: Electrical isolation of pulmonary veins — Device:NaviStar® ThermoCool® Irrigated Tip Ablation Catheter in combination with 3D mapping system CARTO or any future development generations of this product line, provided they are CE marked and the centre has the experience of at least 10 procedures before including a patient into the study.
  Arms: Radiofrequency ablation

SUMMARY:
Comparing efficacy and safety of isolation of the pulmonary veins (PV) using a Cryoballoon catheter versus a radiofrequency ablation with a ThermoCool catheter in patients with paroxysmal atrial fibrillation.

DETAILED DESCRIPTION:
The purpose of this randomized clinical trial is to compare the efficacy and safety of isolating the PVs with either the cryoballoon or a RF ablation technique with a ThermoCool catheter, a system which can be regarded as standard for ablation. In total 762 patients with paroxysmal atrial fibrillation has been randomized for either radiofrequency (RF) or cryoballoon. With both techniques, PV isolation will be performed. Primary end point of the trial is the time to first recurrence of atrial arrhythmias or prescription of anti-arrhythmic drugs after a blanking period of three months. Treatment success will be evaluated by using weekly electrocardiography (ECG) monitoring (transtelephonic transmission/Tele-ECG) and using Holter electrocardiograms.

ELIGIBILITY:
Inclusion Criteria:

* Symptomatic PAF with at least two episodes and at least one episode documented (30 seconds episode length, documented by ECG within last 12 months).
* Documented treatment failure for effectiveness of at least one anti-arrhythmic drug(AAD Type I or III, including β-blocker and AAD intolerance).
* ≥ 18 and ≤ 75 years of age.
* Patients who are mentally and linguistically able to understand the aim of the trial and to show sufficient compliance in following the trial protocol.
* Patient is able to verbally acknowledge and understand the associated risks, benefits, and treatment alternatives to therapeutic options of this trial: cryoballoon ablation system or standard RF ablation technique. The patients, by providing informed consent, agree to these risks and benefits as stated in the patient informed consent document. All the details have been presented to him and he has signed the informed consent form for the trial.

Exclusion Criteria:

General exclusion criteria

* Any disease that limits life expectancy to less than one year.
* Participation in another clinical trial (of a drug, device or biologic), either within the past two months or ongoing.
* Pregnant women or women of childbearing potential not on adequate birth control: only women with a highly effective method of contraception [oral contraception or intrauterine device (IUD)] or sterile women can be randomized.
* Breastfeeding women.
* Substance misuse.
* Active systemic infection.
* Cryoglobulinaemia.
* Previous participation in this clinical trial.
* Employment by the sponsor or by the department of any of the investigators.
* Close relatives of any of the investigators.

Exclusion criteria related to a cardiac condition

* Patients with prosthetic valves.
* Any previous LA ablation or surgery.
* Any cardiac surgery or percutaneous coronary intervention (PCI) within three months prior to enrollment.
* Unstable angina pectoris.
* Myocardial infarction within three months prior to enrollment.
* Symptomatic carotid stenosis.
* Chronic obstructive pulmonary disease with detected pulmonary hypertension.
* Any condition contraindicating chronic anticoagulation.
* Stroke or transient ischemic attack within six months prior to enrollment.
* Any significant congenital heart defect corrected or not (including atrial septal defects or PV abnormalities) but not including patent foramen ovale.
* New York Heart Association (NYHA) class III or IV congestive heart failure.
* EF < 35 % (determined by echocardiography within 60 days of enrollment as documented in patient medical history).
* Anteroposterior LA diameter > 55 mm (by trans-thoracic echocardiography (TTE or TEE) within three months to prior enrollment).
* LA thrombus (TEE diagnostic performed on admission).
* Intracardiac thrombus.
* PV diameter > 26 mm in right sided PVs.
* Mitral prosthesis.
* Hypertrophic cardiomyopathy (see Appendix IX)
* 2° (Type II) or 3° atrioventricular block.
* Brugada syndrome or long QT syndrome.
* Arrhythmogenic right ventricular dysplasia.
* Sarcoidosis.
* PV stent.
* Myxoma.

Exclusion criteria based on laboratory abnormalities

* Thrombocytosis (platelet count > 600,000 / µl), thrombocytopenia (platelet count < 100,000 / µl).
* Any untreated or uncontrolled hyperthyroidism or hypothyroidism.
* Severe renal dysfunction (stage V, requiring or almost requiring dialysis, glomerular filtration rate (GFR) < 15 ml / min).

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 769 (Actual)
Dates: Start 2011-12; Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Karl-Heinz Kuck, Prof. Dr., Principal Investigator — Asklepios Klinikum St. Georg
Locations (19):
- Na Homolce Hospital, Cardiology, Prague, Czechia
- France (4):
  - Hospital Henri Mondor CHU, Service de Cardiologie, Créteil
  - CHU Lyon, Départment de Rythmologie, Hospital Cardiologique Pradel, Lyon
  - Centre Chirurgical Ambroise Paré, Neuilly-sur-Seine
  - La Clinique Pasteur, 45 Avenue de Lombez, Toulouse
- Germany (6):
  - Herz-Zentrum Bad Krozingen, Bad Krozingen
  - Klinik für Kardiologie II mit interventioneller Elektrophysiologie, Bad Neustadt/Saale
  - Cardioangiologisches Centrum Bethanien - CCB, Frankfurt
  - Universitätsklinikum Greifswald Elektrophysiologie, Greifswald
  - Asklepios Klinik St. Georg, Hamburg
  - Herz-Zentrum-Bodensee Konstanz, Konstanz
- Semmelweis University of Medicine, Kardiovaskuläres Zentrum, Budapest, Hungary
- Cardiac Arrhythmia Research Centre Department of Cardiovascular Medicine Centro Cardiologico Monzino University of Milan, Milan, Italy
- Isala Klinieken loc. Weezenlanden Diagram Clinical Resarch, Zwolle, Netherlands
- Spain (4):
  - Hospital Clinic, University of Barcelona, Barcelona
  - Arrhythmia Unit Hospital Clinico San Carlos, Madrid
  - Hospital Universitario Virgen de la Victoria, Department of Cardiology, Campus Teatinos sn, Málaga
  - Hospital Clinico Universtitario, Cardiology Department Arrhythmia Unit, Valencia
- Universitätsspital Basel, Elektrophysiologie/ Kardiologie, Basel, Switzerland

REFERENCES:
- [Background] Furnkranz A, Brugada J, Albenque JP, Tondo C, Bestehorn K, Wegscheider K, Ouyang F, Kuck KH. Rationale and Design of FIRE AND ICE: A multicenter randomized trial comparing efficacy and safety of pulmonary vein isolation using a cryoballoon versus radiofrequency ablation with 3D-reconstruction. J Cardiovasc Electrophysiol. 2014 Dec;25(12):1314-20. doi: 10.1111/jce.12529. Epub 2014 Nov 12. PMID 25146732
- [Result] Kuck KH, Brugada J, Furnkranz A, Metzner A, Ouyang F, Chun KR, Elvan A, Arentz T, Bestehorn K, Pocock SJ, Albenque JP, Tondo C; FIRE AND ICE Investigators. Cryoballoon or Radiofrequency Ablation for Paroxysmal Atrial Fibrillation. N Engl J Med. 2016 Jun 9;374(23):2235-45. doi: 10.1056/NEJMoa1602014. Epub 2016 Apr 4. PMID 27042964
- [Derived] Huang C, Wang J, He C, Yang K, Zhao H, Chen J, Su L. The Efficacy and Safety of Cryoballoon Versus Radiofrequency Ablation for the Treatment of Atrial Fibrillation: A Meta-Analysis of 15 International Randomized Trials. Cardiol Rev. 2024 Nov-Dec 01;32(6):546-553. doi: 10.1097/CRD.0000000000000531. Epub 2024 Oct 4. PMID 37071112
- [Derived] Kuck KH, Brugada J, Furnkranz A, Chun KRJ, Metzner A, Ouyang F, Schluter M, Elvan A, Braegelmann KM, Kueffer FJ, Arentz T, Albenque JP, Kuhne M, Sticherling C, Tondo C; FIRE AND ICE Investigators. Impact of Female Sex on Clinical Outcomes in the FIRE AND ICE Trial of Catheter Ablation for Atrial Fibrillation. Circ Arrhythm Electrophysiol. 2018 May;11(5):e006204. doi: 10.1161/CIRCEP.118.006204. PMID 29700058
- [Derived] Chun KRJ, Brugada J, Elvan A, Geller L, Busch M, Barrera A, Schilling RJ, Reynolds MR, Hokanson RB, Holbrook R, Brown B, Schluter M, Kuck KH; FIRE AND ICE Investigators. The Impact of Cryoballoon Versus Radiofrequency Ablation for Paroxysmal Atrial Fibrillation on Healthcare Utilization and Costs: An Economic Analysis From the FIRE AND ICE Trial. J Am Heart Assoc. 2017 Jul 27;6(8):e006043. doi: 10.1161/JAHA.117.006043. PMID 28751544
- [Derived] Kuck KH, Furnkranz A, Chun KR, Metzner A, Ouyang F, Schluter M, Elvan A, Lim HW, Kueffer FJ, Arentz T, Albenque JP, Tondo C, Kuhne M, Sticherling C, Brugada J; FIRE AND ICE Investigators. Cryoballoon or radiofrequency ablation for symptomatic paroxysmal atrial fibrillation: reintervention, rehospitalization, and quality-of-life outcomes in the FIRE AND ICE trial. Eur Heart J. 2016 Oct 7;37(38):2858-2865. doi: 10.1093/eurheartj/ehw285. Epub 2016 Jul 5. PMID 27381589
- [Derived] Luik A, Radzewitz A, Kieser M, Walter M, Bramlage P, Hormann P, Schmidt K, Horn N, Brinkmeier-Theofanopoulou M, Kunzmann K, Riexinger T, Schymik G, Merkel M, Schmitt C. Cryoballoon Versus Open Irrigated Radiofrequency Ablation in Patients With Paroxysmal Atrial Fibrillation: The Prospective, Randomized, Controlled, Noninferiority FreezeAF Study. Circulation. 2015 Oct 6;132(14):1311-9. doi: 10.1161/CIRCULATIONAHA.115.016871. Epub 2015 Aug 17. PMID 26283655
- See also: Rationale and Design of FIRE AND ICE: A Multicenter Randomized Trial Comparing Efficacy and Safety of Pulmonary Vein Isolation using a Cryoballoon Versus Radiofrequency Ablation with 3D-reconstruction. — http://www.ncbi.nlm.nih.gov/pubmed/25146732
- See also: Cryoballoon or Radiofrequency Ablation for Paroxysmal Atrial Fibrillation. — http://www.ncbi.nlm.nih.gov/pubmed/27042964
- See also: FIRE AND ICE: LBCT ACC — http://www.acc.org/latest-in-cardiology/clinical-trials/2016/04/03/15/28/fire-and-ice

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 769 subjects were enrolled; 7 subjects exited prior to randomization, 762 were randomized
Period: Overall Study
Arm/Group | Cryoballoon Ablation | Radiofrequency Ablation
Started | 378 (378 subjects randomized to Cryoballoon arm) | 384 (384 subjects randomized to radiofrequency arm)
Completed | 374 (374 received ablation) | 376 (376 received ablation)
Not Completed | 4 | 8
Not completed — Inclusion/Exclusion Criteria Violation | 3 | 3
Not completed — Physician Decision | 1 | 0
Not completed — Withdrawal by Subject | 0 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cryoballoon Ablation | Radiofrequency Ablation | Total
Number analyzed (Participants) | 374 | 376 | 750
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.9 (9.8) | 60.1 (9.2) | 60.0 (9.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 153 | 140 | 293
  Male | 221 | 236 | 457
Years since first PAF diagnosis [Mean (Standard Deviation); unit: years] | 4.6 (5.1) | 4.7 (5.3) | 4.6 (5.2)

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects With Recurrence of Atrial Arrhythmias or Prescription of Anti-arrhythmic Drug or Re-ablation After a Blanking Period of Three Months After the Initial Ablation Procedure
Description: Number of subjects reporting a primary efficacy endpoint
Time Frame: 33 months
Population: Subjects randomized and received an ablation procedure. Modified intent-to-treat (mITT) population.
Measure: Count of Participants; unit: Participants
Arm/Group | Cryoballoon Ablation | Radiofrequency Ablation
Number analyzed (Participants) | 374 | 376
Participants | 138 | 143

2. Primary Outcome: Number of Subjects With a Primary Safety Event. A Primary Safety Event Includes a Composite of Death (Including Cardiovascular Death), All-cause Stroke/Transient Ischemic Attack (TIA) and Serious Adverse Events of Special Interest.
Time Frame: 33 months
Population: Subjects randomized and received an ablation procedure. Modified intent-to-treat (mITT) population.
Measure: Count of Participants; unit: Participants
Arm/Group | Cryoballoon Ablation | Radiofrequency Ablation
Number analyzed (Participants) | 374 | 376
Participants
  No primary safety event | 334 | 325
  Death | 2 | 0
  All-cause stroke or TIA | 2 | 2
  Atrial Arrhythmia | 8 | 13
  Non-arrhythmia-related Serious Adverse Event | 28 | 36

3. Secondary Outcome: All-cause Death
Time Frame: 33 months
Population: Subjects randomized and received ablation. Modified intent-to-treat (mITT) population.
Measure: Count of Participants; unit: Participants
Arm/Group | Cryoballoon Ablation | Radiofrequency Ablation
Number analyzed (Participants) | 374 | 376
Participants | 2 | 0

4. Secondary Outcome: Arrhythmia-related Death
Time Frame: 33 months
Population: Subjects randomized and received an ablation procedure. Modified intent-to-treat (mITT) population.
Measure: Count of Participants; unit: Participants
Arm/Group | Cryoballoon Ablation | Radiofrequency Ablation
Number analyzed (Participants) | 374 | 376
Participants | 0 | 0

5. Secondary Outcome: Total Procedure Duration
Time Frame: Through the initial ablation procedure
Population: Subjects randomized and received ablation. Modified intent-to-treat (mITT) population.
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Cryoballoon Ablation | Radiofrequency Ablation
Number analyzed (Participants) | 374 | 376
minutes | 124.4 (39.0) | 140.9 (54.9)

6. Secondary Outcome: Total Time of Fluoroscopy
Time Frame: Fluoroscopy meter time through the initial ablation procedure
Population: Subjects randomized and received ablation procedure. Modified intent-to-treat (mITT) population
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Cryoballoon Ablation | Radiofrequency Ablation
Number analyzed (Participants) | 374 | 376
minutes | 16.6 (17.8) | 21.7 (13.9)

7. Secondary Outcome: Number of Subjects Reporting a Cardiovascular Hospitalization Over the Duration of the Study.
Time Frame: 33 months
Population: Subjects randomized and received an ablation procedure. Modified intent-to-treat (mITT) population.
Measure: Count of Participants; unit: Participants
Arm/Group | Cryoballoon Ablation | Radiofrequency Ablation
Number analyzed (Participants) | 374 | 376
Participants | 89 | 135

8. Secondary Outcome: Number of Cardiovascular Hospitalizations
Description: The total number of cardiovascular hospitalizations reported over the duration of the study.
Time Frame: 33 months
Population: Subjects randomized and received an ablation procedure. Modified intent-to-treat (mITT) population.
Measure: Number; unit: number of cardiovascular hospitalization
Arm/Group | Cryoballoon Ablation | Radiofrequency Ablation
Number analyzed (Participants) | 374 | 376
number of cardiovascular hospitalization | 139 | 203

ADVERSE EVENTS:
Time Frame: The duration of the study. Mean follow-up was 1.5 years, maximum follow-up was 33 months.
Arm/Group | Cryoballoon Ablation | Radiofrequency Ablation
Serious Adverse Events (participants affected / at risk) | 129/374 | 158/376
Other Adverse Events (participants affected / at risk) | 0/374 | 0/376
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cryoballoon Ablation (N=374) | Radiofrequency Ablation (N=376)
ABDOMINAL PAIN UPPER (Gastrointestinal disorders) | 2 (2) | 0 (0)
ACCIDENT (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
ADVERSE DRUG REACTION (General disorders) | 0 (0) | 1 (1)
ANESTHETIC COMPLICATION PULMONARY (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
ANGINA PECTORIS (Cardiac disorders) | 1 (1) | 0 (0)
ANGINA UNSTABLE (Cardiac disorders) | 1 (1) | 0 (0)
ANXIETY (Psychiatric disorders) | 1 (1) | 0 (0)
AORTIC ANEURYSM (Vascular disorders) | 1 (1) | 1 (1)
AORTIC DISSECTION (Vascular disorders) | 1 (2) | 0 (0)
ARTERIOGRAM CORONARY (Investigations) | 0 (0) | 1 (1)
ARTERIOVENOUS FISTULA (Vascular disorders) | 0 (0) | 3 (3)
ARTERITIS (Vascular disorders) | 1 (1) | 0 (0)
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
ASPIRATION (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
ASTHENIA (General disorders) | 2 (2) | 2 (2)
ATRIAL FIBRILLATION (Cardiac disorders) | 54 (69) | 86 (110)
ATRIAL FLUTTER (Cardiac disorders) | 8 (10) | 12 (13)
ATRIAL SEPTAL DEFECT (Congenital, familial and genetic disorders) | 1 (2) | 0 (0)
ATRIAL TACHYCARDIA (Cardiac disorders) | 5 (6) | 7 (7)
ATRIOVENTRICULAR BLOCK SECOND DEGREE (Cardiac disorders) | 0 (0) | 1 (1)
BENIGN PROSTATIC HYPERPLASIA (Reproductive system and breast disorders) | 0 (0) | 2 (2)
BENIGN SALIVARY GLAND NEOPLASM (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
BILIARY COLIC (Hepatobiliary disorders) | 0 (0) | 1 (1)
BRACHYTHERAPY TO UTERUS (Surgical and medical procedures) | 1 (1) | 0 (0)
BRADYCARDIA (Cardiac disorders) | 0 (0) | 1 (1)
BREAST CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
BRONCHIAL NEOPLASM BENIGN (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
BRONCHITIS (Infections and infestations) | 1 (1) | 1 (1)
BURSITIS (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
CARCINOID TUMOUR OF THE CAECUM (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
CARDIAC ABLATION (Surgical and medical procedures) | 1 (1) | 1 (1)
CARDIAC FAILURE (Cardiac disorders) | 0 (0) | 1 (1)
CARDIAC TAMPONADE (Cardiac disorders) | 1 (1) | 4 (4)
CEREBELLAR INFARCTION (Nervous system disorders) | 0 (0) | 1 (1)
CEREBRAL HEMORRHAGE (Nervous system disorders) | 0 (0) | 1 (1)
CERVICAL VERTEBRAL FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
CHEST PAIN (General disorders) | 0 (0) | 1 (1)
CHOKING (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
CHOLECYSTECTOMY (Surgical and medical procedures) | 0 (0) | 1 (1)
CHOLECYSTITIS (Hepatobiliary disorders) | 1 (1) | 1 (1)
CHOLELITHIASIS (Hepatobiliary disorders) | 0 (0) | 1 (1)
CHRONIC OBSTRUCTIVE PULMONARY DISEASE (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
CIRCULATORY COLLAPSE (Vascular disorders) | 1 (1) | 0 (0)
CONTRAST MEDIA REACTION (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
CONTUSION (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
CORONARY ARTERY DISEASE (Cardiac disorders) | 1 (1) | 2 (2)
CORONARY ARTERY STENOSIS (Cardiac disorders) | 1 (1) | 0 (0)
CRITICAL ILLNESS POLYNEUROPATHY (Nervous system disorders) | 1 (1) | 0 (0)
DACRYOSTENOSIS ACQUIRED (Eye disorders) | 1 (1) | 0 (0)
DEATH (General disorders) | 1 (1) | 0 (0)
DEVICE RELATED INFECTION (Infections and infestations) | 0 (0) | 1 (1)
DIABETIC GASTROPARESIS (Gastrointestinal disorders) | 1 (1) | 0 (0)
DIARRHOEA (Gastrointestinal disorders) | 1 (1) | 0 (0)
DISSOCIATIVE DISORDER (Psychiatric disorders) | 1 (1) | 0 (0)
DIVERTICULITIS (Infections and infestations) | 2 (3) | 0 (0)
DIZZINESS (Nervous system disorders) | 1 (1) | 4 (4)
DYSARTHRIA (Nervous system disorders) | 1 (1) | 0 (0)
DYSPNEA (Respiratory, thoracic and mediastinal disorders) | 7 (7) | 4 (4)
DYSPNEA EXERTIONAL (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
DYSURIA (Renal and urinary disorders) | 0 (0) | 1 (1)
ENTEROCOLITIS (Gastrointestinal disorders) | 1 (1) | 0 (0)
EPIGASTRIC DISCOMFORT (Gastrointestinal disorders) | 0 (0) | 1 (1)
EPILEPSY (Nervous system disorders) | 1 (1) | 0 (0)
EXERTIONAL DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
EXOSTOSIS OF EXTERNAL EAR CANAL (Ear and labyrinth disorders) | 1 (1) | 0 (0)
FACIAL BONES FRACTURE (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
FATIGUE (General disorders) | 1 (1) | 0 (0)
FEMORAL NECK FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
GASTRITIS (Gastrointestinal disorders) | 0 (0) | 2 (2)
GASTROINTESTINAL HEMORRHAGE (Gastrointestinal disorders) | 0 (0) | 1 (1)
GROIN PAIN (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
HEMATOCHEZIA (Gastrointestinal disorders) | 0 (0) | 1 (1)
HEMATOMA (Vascular disorders) | 2 (2) | 5 (6)
HEMATOMA EVACUATION (Surgical and medical procedures) | 0 (0) | 1 (1)
HEMATURIA (Renal and urinary disorders) | 0 (0) | 1 (1)
HEMOPTYSIS (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
HEMORRHAGE (Vascular disorders) | 4 (4) | 0 (0)
HERNIA (General disorders) | 1 (1) | 0 (0)
HODGKIN'S DISEASE (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
HOSPITALISATION (Surgical and medical procedures) | 0 (0) | 1 (1)
HYPERHIDROSIS (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
HYPERTENSION (Vascular disorders) | 2 (3) | 2 (2)
HYPERTENSIVE CRISIS (Vascular disorders) | 1 (1) | 0 (0)
HYPERTENSIVE ENCEPHALOPATHY (Nervous system disorders) | 1 (1) | 0 (0)
HYPOAESTHESIA (Nervous system disorders) | 0 (0) | 1 (1)
HYPONATREMIA (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
HYSTEROSALPINGO-OOPHORECTOMY (Surgical and medical procedures) | 1 (1) | 0 (0)
IMPAIRED GASTRIC EMPTYING (Gastrointestinal disorders) | 1 (1) | 0 (0)
INFECTIVE EXACERBATION OF CHRONIC OBSTRUCTIVE AIRWAYS DISEASE (Infections and infestations) | 0 (0) | 1 (2)
INTESTINAL PERFORATION (Gastrointestinal disorders) | 1 (1) | 0 (0)
LARGE INTESTINE POLYP (Gastrointestinal disorders) | 0 (0) | 1 (1)
LIP AND/OR ORAL CAVITY CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (2) | 0 (0)
LOCAL SWELLING (General disorders) | 0 (0) | 1 (1)
MENIERE'S DISEASE (Ear and labyrinth disorders) | 0 (0) | 1 (1)
METASTATIC NEOPLASM (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
MICROLITHIASIS (General disorders) | 1 (1) | 0 (0)
MIGRAINE WITH AURA (Nervous system disorders) | 0 (0) | 1 (1)
MULTIPLE SCLEROSIS (Nervous system disorders) | 1 (1) | 0 (0)
MYOCARDIAL INFARCTION (Cardiac disorders) | 0 (0) | 1 (1)
NAUSEA (Gastrointestinal disorders) | 1 (1) | 1 (1)
NEPHROLITHIASIS (Renal and urinary disorders) | 0 (0) | 1 (1)
NODAL OSTEOARTHRITIS (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
OESOPHAGEAL ULCER (Gastrointestinal disorders) | 1 (1) | 0 (0)
OPTIC NEURITIS (Nervous system disorders) | 0 (0) | 1 (1)
OSTEOARTHRITIS (Musculoskeletal and connective tissue disorders) | 2 (2) | 5 (5)
PAIN (General disorders) | 0 (0) | 1 (1)
PAINFUL RESPIRATION (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
PALPITATIONS (Cardiac disorders) | 4 (4) | 9 (11)
PANCREATIC CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
PARAPARESIS (Nervous system disorders) | 1 (1) | 0 (0)
PERICARDIAL EFFUSION (Cardiac disorders) | 1 (1) | 2 (2)
PERICARDITIS (Cardiac disorders) | 1 (1) | 1 (1)
PHARYNGEAL INFLAMMATION (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
PHRENIC NERVE PARALYSIS (Nervous system disorders) | 10 (10) | 0 (0)
PNEUMONIA (Infections and infestations) | 4 (5) | 3 (3)
PNEUMOTHORAX (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
POST PROCEDURAL COMPLICATION (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
POST PROCEDURAL HEMATOMA (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
POST PROCEDURAL HEMORRHAGE (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
POST PROCEDURAL STROKE (Nervous system disorders) | 1 (1) | 0 (0)
PRESYNCOPE (Nervous system disorders) | 2 (2) | 3 (3)
PROCEDURAL DIZZINESS (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
PSORIASIS (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
PULMONARY CONGESTION (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
PULMONARY EMBOLISM (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
PULMONARY OEDEMA (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
PYREXIA (General disorders) | 0 (0) | 2 (2)
RADIUS FRACTURE (Injury, poisoning and procedural complications) | 2 (3) | 0 (0)
RECTAL LESION EXCISION (Surgical and medical procedures) | 1 (1) | 0 (0)
RENAL COLIC (Renal and urinary disorders) | 0 (0) | 1 (1)
RENAL FAILURE ACUTE (Renal and urinary disorders) | 1 (1) | 0 (0)
RESPIRATORY FAILURE (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
RESPIRATORY TRACT INFECTION (Infections and infestations) | 1 (1) | 1 (1)
ROAD TRAFFIC ACCIDENT (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
ROTATOR CUFF SYNDROME (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
SEPSIS (Infections and infestations) | 1 (1) | 0 (0)
SICK SINUS SYNDROME (Cardiac disorders) | 2 (2) | 1 (1)
SJOGREN'S SYNDROME (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
SPINAL COLUMN INJURY (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
SPINAL FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
SPONTANEOUS HEMATOMA (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
STASIS SYNDROME (Gastrointestinal disorders) | 1 (1) | 0 (0)
SUPRAVENTRICULAR EXTRASYSTOLES (Cardiac disorders) | 1 (1) | 2 (2)
SYNCOPE (Nervous system disorders) | 2 (2) | 0 (0)
SYNOVITIS (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
TACHYCARDIA (Cardiac disorders) | 2 (2) | 2 (2)
TENDON RUPTURE (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
THORACOTOMY (Surgical and medical procedures) | 1 (1) | 0 (0)
THYROID CYST (Endocrine disorders) | 0 (0) | 1 (1)
THYROID DISORDER (Endocrine disorders) | 1 (1) | 0 (0)
THYROID NODULE (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
TONSILLECTOMY (Surgical and medical procedures) | 0 (0) | 1 (1)
TONSILLITIS (Infections and infestations) | 0 (0) | 1 (1)
TOXIC NODULAR GOITRE (Endocrine disorders) | 1 (1) | 0 (0)
TRANSIENT GLOBAL AMNESIA (Nervous system disorders) | 0 (0) | 1 (1)
TRANSIENT ISCHEMIC ATTACK (Nervous system disorders) | 1 (1) | 2 (2)
URINARY BLADDER HEMORRHAGE (Renal and urinary disorders) | 0 (0) | 1 (1)
URINARY TRACT INFECTION (Infections and infestations) | 0 (0) | 1 (1)
UTERINE PROLAPSE (Reproductive system and breast disorders) | 0 (0) | 1 (1)
VAGINAL HEMORRHAGE (Reproductive system and breast disorders) | 0 (0) | 1 (1)
VARICOSE VEIN (Vascular disorders) | 1 (1) | 1 (1)
VARICOSE VEIN OPERATION (Surgical and medical procedures) | 0 (0) | 1 (1)
VASCULAR PSEUDOANEURYSM (Injury, poisoning and procedural complications) | 2 (2) | 8 (8)
VASCULITIS (Vascular disorders) | 1 (1) | 0 (0)
VENTRICULAR FIBRILLATION (Cardiac disorders) | 0 (0) | 1 (1)
VENTRICULAR TACHYCARDIA (Cardiac disorders) | 1 (1) | 0 (0)
VESSEL PERFORATION (Vascular disorders) | 0 (0) | 1 (1)
VISUAL IMPAIRMENT (Eye disorders) | 1 (1) | 1 (1)
VOMITING (Gastrointestinal disorders) | 3 (3) | 1 (1)
WOUND INFECTION (Infections and infestations) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less